CLINICAL TRIAL: NCT03598153
Title: A Registry Study of Shujinjianyao Pill Used in Clinical Real World
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy director, China Academy of Chinese Medical Sciences
Other Study IDs: Shujin
Record Dates: First submitted 2018-06-24; First posted 2018-07-26 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-06

CONDITIONS: Sciatica
Keywords: Waist and knee pain; sciatica
MeSH Terms: conditions — Sciatica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Shujinjianyao Pill — According to the usage and dosage of the instructions, patients should use the medicine dialectically and rationally for 4 weeks.

SUMMARY:
The purpose of this study is to get to know how Shujinjianyao Pill in hospital results in drug-induced liver injury or other adverse drug reactions from a cohort event monitoring as registration research.

DETAILED DESCRIPTION:
In order to monitor drug-induced liver injury or other adverse drug reactions of Shujinjianyao Pill in clinical real world, registry study is a suitable method in this area. Meanwhile, the investigators will use nested case-control study to find out the mechanism of drug-induced liver injury. Calculate the incidence of drug-induced liver injury or other adverse drug reactions is one of the main aims for this study. Therefore, Safety monitoring of Shujinjianyao Pill is an very important problem that needs to be done through a large sample observational study. According to the relevant regulations of the state drug administration(SDA), 3000 cases need to be registered at least. The aim population is who use Shujinjianyao Pill with normal liver function before medication from June 2018 to October 2019.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with normal liver function before medication.
* 2.Patients suffered from Waist and knee pain or sciatica.

Exclusion Criteria:

* 1.Patients who are pregnant, phrenetic, and suffered from serious illness.
* 2.Patients suffered from viral hepatitis or autoimmune hepatitis or alcoholic hepatitis or hereditary metabolic hepatitis or cirrhosis or cancer of the liver.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: With normal liver function before medication, patients suffered from waist and knee pain or sciatica.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-07-25 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Is there any abnormality in liver function test index（ALT、AST、TBil、GGT） after using Shujinjianyao Pill about four weeks ? | After using Shujinjianyao Pill about four weeks.
  The liver function test index mainly includes glutamic-pyruvic transaminase(ALT),glutamic-oxalacetic transaminase(AST), gamma-glutamyl transpeptidase(GGT) and total bilirubin(TBil). If the index is abnormal, it indicates abnormal liver function, and severe cases can lead to liver injury.

SECONDARY OUTCOMES:
Is there any abnormality in renal function test index（Bun、Cr） after medication? | After using Shujinjianyao Pill around four weeks.
  The renal function test index mainly includes creatinine(Cr) and urea nitrogen (Bun).
  If the index is abnormal, it indicates abnormal kidney function. We plan to monitor whether medication is harmful to renal function test index.
Is there any abnormality in electrocardiogram after medication? | After using Shujinjianyao Pill around four weeks.
  Electrocardiogram is a special device that amplifies the electrical effects of heart contractions and diastasis by drawing wavy stripes on paper.The observation of electrocardiogram can help diagnose various heart diseases.If someone has an electrocardiogram, doctors use special equipment to measure the electric currents produced by that person's heart in order to see whether it is working normally.
  We want to monitor whether medication is harmful to electrocardiogram.
Is there any abnormality in blood routine examination after medication? | After using Shujinjianyao Pill around four weeks.
  Blood routine examination is a commonly used index for observing the therapeutic effect and guiding medication and treatment.
Is there any abnormality in routine urinalysis after medication? | After using Shujinjianyao Pill around four weeks.
  As an indicator of excretion, routine urinalysis reflects the body's metabolic state and is an important indicator of many diseases.
  We want to monitor whether medication is harmful to routine urinalysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yanming Xie, BA, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui X, Liang L, Wang L, Wang Z, Li Y, Gao Y, Zhang C, Sun M, Wang S, Liu J, Zhang Y, Wang Z, Wei X, Xie Y. Safety of Shujinjianyao pill in clinical real world: A prospective, observational, multicenter, large-sample study Protocol. Medicine (Baltimore). 2019 Aug;98(33):e16853. doi: 10.1097/MD.0000000000016853. PMID 31415416